CLINICAL TRIAL: NCT04548414
Title: The Effect of Homocysteine on the Prognosis of Patients With sepsis-an Observational Study
Brief Title: Homocysteine in Patients With Sepsis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanjing University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jun Lu, MD, Doctor, Nanjing University of Traditional Chinese Medicine
Other Study IDs: aztec04030910
Record Dates: First submitted 2020-09-10; First posted 2020-09-14 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sepsis group: The patients in this group are diagnosed sepsis with the sepsis 3.0 definition.
  Interventions: Other: No.
- Control group: The recruited volunteers in this group are healthy.

INTERVENTIONS:
Other: No. — This is an observational study with no intervention.
  Groups: Sepsis group

SUMMARY:
After stimulation by lipopolysaccharide (LPS), the one-carbon metabolism of macrophages was significantly up-regulated, the expression of key enzyme 5,10-methylenetetrahydrofolate reductase increased. In vitro experiments we found that LPS stimulation can increase the expression of MTHFR mRNA and protein in macrophages, suggesting that aerobic glycolysis may trigger cytokine storm through one-carbon metabolism. Homocysteine (homocysteine, Hcy) is an important intermediate product of one-carbon metabolism. A number of studies have shown that Hcy is positively correlated with the level of pro-inflammatory factors, significantly enhancing cytokine storm. However, the relationship between Hcy and serum pro-inflammatory factors in patients with sepsis and the effect of Hcy on the prognosis of patients with sepsis are still unclear. Based on the previous work, our research group intends to carry out single-center, prospective, observational clinical research to observe the relationship between homocysteine and the mortality of patients with sepsis, and to provide new indicators for accurately judging the prognosis of sepsis , To provide new targets for clinical development of drugs for the treatment of sepsis.

ELIGIBILITY:
Inclusion Criteria:

Patients with sepsis and the age limits between 18-80 years.

Exclusion Criteria:

* Non-septic patients with hyperhomocysteinemia caused by various reasons. ②After the onset, other medicines for the treatment of folate deficiency and hyperhomocysteinemia have been used. ③Women during pregnancy and lactation. ④ Suspected or did have a history of alcohol or drug abuse. ⑤Patients who are participating in clinical trials of other drugs.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patients with sepsis and volunteers who are healthy.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-09-20 (Estimated); Primary Completion 2022-05-19 (Estimated); Study Completion 2022-09-19 (Estimated)

PRIMARY OUTCOMES:
28-day mortality | one month
  the correlation with the level of Hcy and 28-day mortality